CLINICAL TRIAL: NCT06016920
Title: A Phase 1/2a, Open-label, Dose-finding Trial to Evaluate Safety, Immunogenicity, and Anti-tumor Activity of VB10.16 and Pembrolizumab in Patients with Unresectable Recurrent or Metastatic HPV16-positive Head-Neck Squamous Cell Carcinoma
Brief Title: Safety and Efficacy of VB10.16 and Pembrolizumab in Patients with Head-Neck Squamous Cell Carcinoma
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Nykode Therapeutics ASA (Industry)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: VB-C-03; 2022-503055-26-00 (Other: EU Trial Number); KEYNOTE-E72 (Other: Merck Sharp & Dohme LLC); MK-3475-E72 (Other: Merck Sharp & Dohme LLC)
Record Dates: First submitted 2023-08-24; First posted 2023-08-30 (Actual); Last update posted 2024-12-17 (Actual); Status verified 2024-12

CONDITIONS: HPV Positive Oropharyngeal Squamous Cell Carcinoma; HNSCC
Keywords: Unresectable; recurrent; metastatic; HPV16 positive; PD-L1
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis | interventions — pembrolizumab

STUDY DESIGN:
Intervention Model Description: Dose-finding trial, including a dose escalation phase (phase 1) where participants are allocated sequentially to one of the 3 escalating doses; and a dose expansion phase (phase 2a) where participants are randomized to one of two doses
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Phase1: Dose Escalation: 3 mg VB10.16 + Pembrolizumab (Experimental): 3 mg of VB10.16 via i.m. needle-free injections in the deltoid muscles
  Pembrolizumab will be given as standard of care/ background medication via i.v. infusions
  Interventions: Biological: VB10.16; Drug: Pembrolizumab
- Phase 1: Dose Escalation: 6 mg VB10.16 + Pembrolizumab (Experimental): 6 mg of VB10.16 via i.m. needle-free injections in the deltoid muscles and quadriceps or gluteus muscles
  Pembrolizumab will be given as standard of care/ background medication via i.v. infusions
  Interventions: Biological: VB10.16; Drug: Pembrolizumab
- Phase 1: Dose Escalation: 9 mg VB10.16 + Pembrolizumab (Experimental): 9 mg of VB10.16 via i.m. needle-free injections in the deltoid muscles and quadriceps and/or gluteus muscle
  Pembrolizumab will be given as standard of care/ background medication via i.v. infusions
  Interventions: Biological: VB10.16; Drug: Pembrolizumab
- Phase 2: Dose Expansion: High dose of VB10.16 + Pembrolizumab (Experimental): The highest dose of VB10.16 to be safety-cleared in the escalation phase will be given via i.m. needle-free injections in the deltoid muscles and quadriceps and/or gluteus muscle
  Pembrolizumab will be given as standard of care/ background medication via i.v. infusions
  Interventions: Biological: VB10.16; Drug: Pembrolizumab
- Phase 2: Dose Expansion: 3 mg VB10.16 + Pembrolizumab (Experimental): 3 mg of VB10.16 via i.m. needle-free injections in the deltoid muscles
  Pembrolizumab will be given as standard of care/ background medication via i.v. infusions
  Interventions: Biological: VB10.16; Drug: Pembrolizumab

INTERVENTIONS:
Biological: VB10.16 — Intramuscular (i.m.) administrations of VB10.16 every 3 weeks (Q3W) starting at Week 1/Day 1 during a 12-week induction period, followed by a maintenance period with administrations every 6 weeks (Q6W) from Week 13 until Week 48. A total of up to 10 i.m. administrations will be given.
  VB10.16 will be administered via Pharma Jet® Stratis 0.5 mL needle free injection system.
Drug: Pembrolizumab — Pembrolizumab 200 mg intravenous (i.v.) will be given in accordance with the local regulatory-approved label Q3W starting at Week 1/Day 1 for as long as the patient tolerates and continues to have clinical benefit from the treatment based on the patient and investigator's decision, up to a maximum of 35 treatments corresponding to approximately 2 years of treatment.
  After 48 weeks of treatment patients can continue on 200 mg Q3W or change to 400 mg Q6W at the discretion of the investigator and after consultation with the sponsor.
  Pembrolizumab will be given by i.v. infusion over 30 minutes.
  Other Names: KEYTRUDA®

SUMMARY:
This is a multi-center study in patients with un-resectable Recurrent or Metastatic HPV16-positive oropharyngeal Head and Neck Squamous Cell Carcinoma (HNSCC). The trial is designed to investigate VB10.16, an investigational therapeutic DNA vaccine in combination with another medicine, pembrolizumab, which is the standard of care for patients with previously untreated metastatic or resectable recurrent PD-L1 positive HNSCC. The study is divided in 2 parts: a phase 1, dose escalation part, testing 3 different doses of VB10.16 in combination with a standard fixed dose of pembrolizumab. The goal of this part is to evaluate the safety and tolerability of the combined treatment and to decide on the dose of VB10.16 to be used in the second part of the trial. In the second part of the trial, a phase 2a, dose expansion part, participants will receive either the highest safe dose of VB10.16 from part 1 or the 3 mg dose both in combination with pembrolizumab. The dose given to each participant will be decided in random.

The trial is designed to define the optimal dose of VB10.16 in combination with pembrolizumab for future clinical studies based on the safety, tolerability and anti-tumor effect data generated.

DETAILED DESCRIPTION:
This phase 1/2a, open-label, dose-finding trial is designed to evaluate the safety, tolerability, immunogenicity, and anti-tumor activity of VB10.16 immunotherapy in patients with HPV16-positive R/M oropharyngeal HNSCC whose tumors express PDL1 (CPS ≥ 1) and who are eligible for pembrolizumab monotherapy as standard of care. The trial is designed to determine the biological optimal dose (BOD) of VB10.16 in combination with a fixed dose of pembrolizumab based on the totality of data (i.e., safety, tolerability, anti-tumor activity, and HPV16 E6/E7specific cellular immune response). The trial consists of 2 consecutive phases with separate patient groups in a seamless trial design: a dose escalation phase (phase 1) and a dose expansion phase (phase 2a). After completing 48 weeks of combination treatment, patients can either continue pembrolizumab treatment with 200 mg Q3W administration or change to 400 mg Q6W administration at the discretion of the investigator and after consultation with the Sponsor.

ELIGIBILITY:
Inclusion Criteria:

GENERAL REQUIREMENTS

1. ≥18 years of age (or as per national legal age of trial consent, whichever is higher) at date of signing the informed consent form (ICF)
2. Histologically or cytologically confirmed R/M HNSCC, located in the oropharynx, considered incurable by local therapy and eligible for monotherapy with pembrolizumab
3. HPV16 positivity of R/M oropharyngeal HNSCC confirmed by designated central laboratory
4. PD-L1 positivity (CPS ≥1) using the validated PD-L1 IHC 22C3 pharmDx (DAKO) assay.
5. Primary tumor location in the oropharynx.
6. At least 1 measurable lesion per RECIST 1.1

   ORGAN FUNCTION

   Overall function:
7. Eastern Cooperative Oncology Group (ECOG) performance status (PS) ≤ 1

   Hematological function:
8. Platelets ≥100 × 10^9/L (100,000/µL)
9. Neutrophils (absolute neutrophil count [ANC]) ≥1.5 × 10^9/L (1,500/µL)
10. Hemoglobin ≥5.6 mmol/L (9.0 g/dL)

    Hepatic and hemostatic function:
11. Bilirubin (BILI), total ≤1.5 × upper limit of normal (ULN) (except Gilbert syndrome, then direct BILI ≤2 × ULN) or direct bilirubin ≤ULN for participants with total bilirubin levels >1.5 × ULN.
12. Aspartate transaminase (AST) ≤ 2.5 × ULN or ≤5 × ULN for a patient with liver metastases.
13. Alanine transaminase (ALT) ≤ 2.5 × ULN or ≤5 × ULN for a patient with liver metastases.
14. Alkaline phosphatase ≤ 2.5 × ULN or ≤5 × ULN for a patient with liver metastases.
15. International normalized ratio (INR) or prothrombin time (PT) ≤1.5 × ULN unless the patient is receiving anticoagulant therapy, in which case PT and partial thromboplastin time (PTT)/activated PTT (aPTT) must be within therapeutic range of intended use of anticoagulants.

    Renal function:
16. Estimated glomerular filtration rate (eGFR) ≥45 mL/min/1.73 m^2 using the Cockroft-Gault formula

    OTHER TRIAL REQUIREMENTS
17. Female patients of childbearing potential: negative serum pregnancy test (≤72 hours)
18. Female patients of childbearing potential must agree to use highly effective contraception throughout the trial (14 days prior to initiation of treatment for oral contraception), and for at least 120 days (according to the current version of the IB for pembrolizumab) after the last dose of pembrolizumab and up to 6 months after the last dose of VB10.16, whichever comes last.

    Male patients must agree to use male condoms during intercourse throughout the trial, and up to 3 months after the last dose of VB10.16, and must refrain from sperm donation in the same period.
19. Patients capable of giving informed consent must provide signed and dated written informed consent prior to initiation of any study-related procedures.

Exclusion Criteria:

HNSCC DISEASE

1. Has disease that is suitable for local therapy with curative intent
2. Has progressive disease ≤6 months after completion of curatively intended concurrent chemoradiotherapy for locoregionally advanced R/M oropharyngeal HNSCC
3. Primary tumor site of the oral cavity, hypopharynx, larynx or nasopharynx (any histology)
4. Rapidly progressing disease (e.g., tumor bleeding, uncontrolled tumor pain) in the opinion of the investigator

   PRIOR, CONCURRENT, OR FUTURE INTERVENTIONS
5. Has received prior palliative radiotherapy within 2 weeks of start of trial treatment or has a prior history of radiation pneumonitis
6. Any prior investigational or approved systemic antineoplastic drug or invasive medical device (including ICIs), either as monotherapy or as part of a combination regimen administered in the R/M HNSCC setting
7. Prior solid organ or tissue transplantation (except corneal transplant)
8. Prior autologous or allogeneic hematopoietic stem cell transplantation (HSCT)
9. Prior chimeric antigen receptor T (CAR-T) cell therapy
10. Prior therapy with a monoclonal or bispecific antibody or antibody fragment (or other molecule with similar mechanism of action) that engages T-cells
11. Has received a live or live-attenuated vaccine within 30 days prior to the first dose of trial intervention
12. Administration of severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2) vaccine within 30 days prior to VB10.16 treatment start
13. Prior administration with a therapeutic HPV16 vaccine
14. Patients receiving systemic immunosuppression with immunosuppressive agents such as cyclosporine, azathioprine, methotrexate, or tumor necrosis factor alpha (TNF α) blockers for any concurrent condition
15. Chronic administration of systemic corticosteroids: prednisone >10 mg daily (or dose equivalent)
16. Administration of G-CSF/GM-CSF or transfusions with red blood cells, platelets, or plasma components ≤2 weeks prior to VB10.16 treatment start
17. Has received prior therapy with an anti-PD-1, anti-PD-L1, or anti-PD-L2 agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (e.g., CTLA-4, OX 40, CD137)
18. Has received prior surgery within 4 weeks prior to treatment
19. Any planned major surgery

    PRIOR OR CONCURRENT MORBIDITY

    Malignancy:
20. Past or current malignancy other than inclusion diagnosis, except for:

    * Malignancy treated with curative intent and with no known active disease present and has not received chemotherapy for at least 3 years before screening and felt to be at low risk for recurrence by the treating physician
    * Adequately treated breast ductal carcinoma in situ without evidence of disease
    * Adequately treated cervical carcinoma in situ, without evidence of disease
    * Adequately treated non-melanoma skin cancer without evidence of disease
    * Adequately treated superficial or in situ carcinoma of the bladder without evidence of disease
    * Prostatic intraepithelial neoplasia without evidence of prostate cancer

    Hepatic and hemostatic function:
21. Any current bleeding disorder, active bleeding, or bleeding diathesis

    Cardiovascular function:
22. Symptomatic congestive heart failure (Grade III or IV as classified by the New York Heart Association), unstable angina pectoris, or cardiac arrhythmia
23. History of myocardial infarction ≤ 6 months prior to planned VB10.16 treatment start
24. Uncontrolled hypertension (systolic blood pressure ≥160 mmHg and/or diastolic blood pressure ≥100 mmHg), despite optimal medical management
25. Any other significant cardiac disease(s) that, in the opinion of the investigator, is/are clinically significant and/or unacceptable

    Pulmonary function:
26. Has a history of (non-infectious) pneumonitis / interstitial lung disease that required steroids or has current pneumonitis / interstitial lung disease

    Immune system and infectious diseases:
27. Primary immunodeficiency, other immunosuppressive disorder, and/or other causes of immunosuppression
28. Has an active autoimmune disease that has required systemic treatment in the past 2 years (i.e., with use of disease-modifying agents, corticosteroids, or immunosuppressive drugs). Replacement therapy (e.g., thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
29. Has a known history of human immunodeficiency virus (HIV) infection.
30. Has a known history of Hepatitis B (defined as HBsAg reactive) or known active Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection
31. Any active, acute, or chronic infection that is uncontrolled and/or requires systemic treatment
32. Known allergies, sensitivity, or intolerance to VB10.16 (active substance or to any of the excipients), pembrolizumab (active substance or to any of the excipients), or aminoglycosides (especially kanamycin).

    Central nervous system (CNS) function:
33. Any history of intracerebral arteriovenous malformations, cerebral aneurysm, or stroke
34. Has known active CNS metastases and/or carcinomatous meningitis. Patients with previously treated brain metastases may participate provided they are radiologically stable, i.e., without evidence of progression for at least 4 weeks by repeat imaging (note that the repeat imaging should be performed during trial screening), clinically stable and without requirement of steroid treatment for at least 14 days prior to first dose of trial treatment
35. New (≤6 months), progressive and/or symptomatic brain metastases

    OTHER
36. Is currently participating in or has participated in a trial of an investigational agent or device in the R/M setting.
37. Has a history or current evidence of any condition, therapy, or laboratory abnormality, or other circumstance that might confound the results of the trial or interfere with the patient's participation for the full duration of the trial, such that it is not in the best interest of the patient to participate, in the opinion of the treating investigator
38. Has a known psychiatric or substance abuse disorder that would interfere with the patient's ability to cooperate with the requirements of the trial
39. Has a concomitant medical condition requiring receipt of a therapeutic anticoagulant that, in the opinion of the treating physician, would contraindicate administration of VB10.16 and tumor biopsies
40. Female patients who are pregnant or breastfeeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Estimated)
Dates: Start 2023-12-19 (Actual); Primary Completion 2027-09 (Estimated); Study Completion 2028-01 (Estimated)

PRIMARY OUTCOMES:
Phase 1: Dose Escalation: Dose Limiting Toxicities (DLT) | 42 days
  Proportion of patient with Dose Limiting Toxicities (DLTs).
Phase 2: Dose Expansion: AEs | 12 months
  Proportion of patients with AEs following treatment initiation by severity grade.
Phase 2: Dose Expansion: Discontinuation due to adverse reaction | 12 months
  Proportion of patients who discontinue due to an adverse reaction.
Phase 2: Dose Expansion: Objective Response Rate (ORR) | 12 months
  Objective Response Rate (ORR), defined as the proportion of patients who have either confirmed CR or confirmed PR as best overall response per RECIST 1.1.
Phase 2: Dose Expansion: Immune response | 12 months
  Change from baseline in HPV16 E6/E7-specific T-cell responses as measured by IFN-γ ELISpot in post-vaccination samples.
Phase 1+2: Full trial: Objective Response Rate (ORR) | 12 months
  Objective Response Rate (ORR), defined as the proportion of patients who have either confirmed CR or confirmed PR as best overall response (BOR) per RECIST 1.1.
Phase 1+2: Full trial: Objective Response Rate (ORR) | 24 months
  Objective Response Rate (ORR), defined as the proportion of patients who have either confirmed CR or confirmed PR as best overall response per RECIST 1.1.

SECONDARY OUTCOMES:
Phase 2: Dose Expansion: Disease control rate (DCR) | 12 months
  Disease control rate (DCR), defined as the proportion of patients who have either confirmed CR, confirmed PR, or SD as BOR according to RECIST 1.1.
Phase 2: Dose Expansion: Duration of response (DOR) | 12 months
  Duration of response (DOR), defined as time from the date of first documented response of CR or PR to the date of the first documented progression or death due to any cause.
Phase 2: Dose Expansion: Duration of response (DOR) | 24 months
  Duration of response (DOR), defined as time from the date of first documented response of CR or PR to the date of the first documented progression or death due to any cause.
Phase 2: Dose Expansion: Duration of complete response (DOCR) | 12 months
  Duration of complete response (DOCR), defined as time from the date of first documented response of CR to the date of the first documented progression or death due to any cause.
Phase 2: Dose Expansion: Duration of Disease Control (DODC) | 12 months
  Duration of Disease Control (DODC), defined as time from the date of first documented response of CR, PR or SD to the date of the first documented progression or death due to any cause.
Phase 2: Dose Expansion: Time to Response (TTR) | 12 months
  Time to Response (TTR), s defined as the time from VB10.16 treatment start date to the date of first documented response of either confirmed CR or confirmed PR.
Phase 2: Dose Expansion: Progression-free survival (PFS) | 12 months
  Progression-free survival (PFS), defined as the time from the VB10.16 treatment start date to the date of the first documented progression or death from any cause, whichever occurs first.
Phase 2: Dose Expansion: Progression-free survival (PFS) | 24 months
  Progression-free survival (PFS), defined as the time from the VB10.16 treatment start date to the date of the first documented progression or death from any cause, whichever occurs first.
Phase 2: Dose Expansion: Overall Survival (OS) | 12 months
  Overall survival (OS), defined as the time from VB10.16 treatment start date to the date of death from any cause.
Phase 2: Dose Expansion: Overall Survival (OS) | 24 months
  Overall survival (OS), defined as the time from VB10.16 treatment start date to the date of death from any cause.
Phase 2: Dose Expansion: Proportion of progression-free | 6 months
  Proportion of patients who are progression-free and alive.
Phase 2: Dose Expansion: Proportion of progression-free | 12 months
  Proportion of patients who are progression-free and alive.
Phase 2: Dose Expansion: Patients alive | 6 months
  Proportion of patients who are alive.
Phase 2: Dose Expansion: Patients alive | 12 months
  Proportion of patients who are alive.
Phase 1+2: Full Trial: Duration of response (DOR) | 12 months
  Duration of response (DOR), defined as time from the date of first documented response of CR or PR to the date of the first documented progression or death due to any cause.
Phase 1+2: Full Trial: Duration of response (DOR) | 24 months
  Duration of response (DOR), defined as time from the date of first documented response of CR or PR to the date of the first documented progression or death due to any cause.
Phase 1+2: Full Trial: Progression-free survival (PFS) | 12 months
  Progression-free survival (PFS), defined as the time from the VB10.16 treatment start date to the date of the first documented progression or death from any cause, whichever occurs first.
Phase 1+2: Full Trial: Progression-free survival (PFS) | 24 months
  Progression-free survival (PFS), defined as the time from the VB10.16 treatment start date to the date of the first documented progression or death from any cause, whichever occurs first.
Phase 1+2: Full Trial: Proportion of progression-free | 12 months
  Proportion of patients who are progression-free and alive.
Phase 1+2: Full Trial: Proportion of progression-free | 24 months
  Proportion of patients who are progression-free and alive.
Phase 1+2: Full Trial: Overall Survival (OS) | 12 months
  Overall survival (OS), defined as the time from VB10.16 treatment start date to the date of death from any cause.
Phase 1+2: Full Trial: Overall Survival (OS) | 24 months
  Overall survival (OS), defined as the time from VB10.16 treatment start date to the date of death from any cause.
Phase 1+2: Full Trial: Patients alive | 12 months
  Proportion of patients who are alive.
Phase 1+2: Full Trial: Patients alive | 24 months
  Proportion of patients who are alive.
Phase 1+2: Full trial: AEs following treatment initiation | 12 months
  Proportion of patients with AEs following treatment initiation by severity grade.
Phase 1+2: Full trial: AEs following treatment initiation | 24 months
  Proportion of patients with AEs following treatment initiation by severity grade.
Phase 1+2: Full Trial: Discontinuation due to an adverse reaction | 12 months
  Proportion of patients who discontinue due to an adverse reaction.
Phase 1+2:Full Trial: Discontinuation due to an adverse reaction | 24 months
  Proportion of patients who discontinue due to an adverse reaction.
Phase 1+2: Full Trial: Immune response | 12 months
  Change from baseline in HPV16 E6/E7-specific T-cell responses as measured by IFN-γ ELISpot in post-vaccination samples.

CONTACTS AND LOCATIONS:
Overall Officials: Åse Bratland, MD, PhD, Principal Investigator — Oslo University Hospital
Locations (17):
- Fakultni nemocnice Olomouc, Olomuoc, Olomouc, Czechia
- France (4):
  - Hôpital de la Pitié - Salpétrière in Paris, Paris, Paris
  - Hospices Civils De Lyon, Lyon
  - CRLC Val d'Aurelle - Institut de Recherche en Cancerologie de Montpellier (IRCM), Montpellier
  - Institut Gustave Roussy, Paris, Paris
- Universität Leipzig Klinik und Poliklinik für Hals-, Nasen-, Ohrenheilkunde, Leipzig, Germany
- Orszagos Onkologiai Intezet, Budapest, Budapest, Hungary
- Norway (2):
  - University of Bergen, Haukeland University Hospital, Bergen
  - Oslo Universitetssykehus, Oslo
- Poland (3):
  - Uniwersyteckie Cetrum Kliniczne, Gdansk
  - Narodowy Instytut Onkologii-im Marii Sklodowskiej-Curie Panstwowy Instytut, Gliwice
  - KO-MED Centra Kliniczne Lublin II, Lublin, Lublin
- Spain (4):
  - Hospital del Mar, Barcelona, Barcelona
  - Institut Catala d'Oncologia, Barcelona, Barcelona
  - Hospital Universitario Virgen de las Nieves, Granada, Granada
  - MD Anderson Cancer Center, Madrid, Madrid
- East and North Hertfordshire NHS Trust Mount Vernon Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No